CLINICAL TRIAL: NCT06229678
Title: Ketones, Muscle Metabolism, and SGLT2 Inhibitors
Brief Title: Ketones, SGLT2, HFrEF
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00000012; R01DK107680 (NIH)
Record Dates: First submitted 2023-12-18; First posted 2024-01-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Type2diabetes; Heart Failure With Reduced Ejection Fraction
Keywords: ketones; cardiovascular benefit
MeSH Terms: conditions — Ketosis | interventions — empagliflozin; Tablets; acipimox

STUDY DESIGN:
Intervention Model Description: A randomized (2:1) placebo controlled double blind study
Who Masked: Participant, Investigator
Masking Description: Participants, and investigators will be blinded to the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin Group (Experimental): Subjects will be randomized 2:1 to receive empagliflozin, 25mg/day for 3 months
  Interventions: Drug: Empagliflozin 25 MG Oral Tablet; Drug: Acipimox 250 Mg Oral Capsule
- Placebo group (Placebo Comparator): Subjects will be randomized to receive the empagliflozin placebo for 3 months
  Interventions: Drug: Placebo; Drug: Acipimox 250 Mg Oral Capsule

INTERVENTIONS:
Drug: Empagliflozin 25 MG Oral Tablet — Empagliflozin 25MG will be administered orally once per day for 3 months
  Other Names: jardiance
  Arms: Empagliflozin Group
Drug: Placebo — The placebo will be administered orally once per day for 3 months
  Arms: Placebo group
Drug: Acipimox 250 Mg Oral Capsule — subjects will be started on acipimox 250mg every 6 hours for 8 days while on continued empagliflozin/placebo therapy. This will be added at the end of 3 months after they finished baseline studies

SUMMARY:
The study team will examine the effects of elevated plasma ketone levels following initiation of SGLT2 inhibitor therapy in high-risk type 2 diabetes mellitus (T2DM) individuals with heart failure (HF) with reduced ejection fraction (HFrEF) providing an energy-rich fuel that is taken up with great avidity by the myocardium, to measure change in Left Ventricle diastolic and systolic function

DETAILED DESCRIPTION:
The study team will examine the effects of elevated plasma ketones caused by 12-week treatment with an SGLT2i (empagliflozin) treatment in participants with T2DM and HF. The study team will focus on three possible mechanisms of action for these effects and test the following:

(i) Skeletal muscle bioenergetics. Using 31P-MRS, the team will quantify phosphocreatine [PCr], ATP, inorganic phosphate, phosphodiester, and intracellular pH. With 1H-MRS, and will measure intramyocellular lipid content at rest and ATPmax production after exercise. The team will examine the relationships between phosphorous metabolite concentrations, intramyocellular lipid content, and ATP generation before and after 12 weeks of SGLT2 inhibition.

(ii) LV systolic and diastolic function using cardiac MRI in type 2 diabetic patients with Class II-III NYHA heart failure and reduced EF.

(iii) To examine the contribution of the SGLT2i-induced increase in plasma ketone concentration on myocardial function and myocardial blood flow by inhibiting the rise in plasma ketone concentration with acipimox while continuing empagliflozin.

(iv) Improvements in Patient-Reported Outcomes (PRO). Kansas City Cardiomyopathy Questionnaire ( KCCQ) scoring will be used to evaluate self-reported physical function and well-being. This tool is a well-developed and validated method to obtain patient self-reported parameters of health in adults.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Class II-III New York Heart Association (NYHA) heart failure and reduced ejection fraction (EF) <50%
* Age 18-80 years
* BMI 23-44 kg/m2
* Glycated hemoglobin (HbA1c) 6.0-10.0%
* Blood Pressure (BP) ≤ 145/85 mmHg
* Estimated glomerular filtration rate (eGFR) ≥30 ml/min•1.73 m2
* Only Type 2 diabetics treated with diet/exercise, metformin, sulfonylureas, metformin/sulfonylurea, Glucagon-like peptide-1 receptor agonist (GLP-1 RA), or insulin
* Stable body weight (±4 pounds) over the previous 3 months prior to enrollment
* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Heart failure due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, severe valvular heart disease, hypertrophic obstructive cardiomyopathy.
* Significant change in diuretic management during the month prior to screening (defined by doubling of diuretic dose or addition of another heart failure medication)
* Type 2 Diabetics treated with Dipeptidyl Peptidase-4 Inhibitor (DPP4i) or pioglitazone
* Pregnancy, lactation, or plans to become pregnant. A negative pregnancy test will be performed before each MRI study to assess current status. For women of child-bearing age (WOCBA) willingness to use contraception, if applicable.
* Allergy/sensitivity to study drugs or their ingredients.
* Cancer.
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Phosphocreatine | Baseline to 3 months
  A measure of phosphocreatine change from baseline to study end
Change in Adenosine Triphosphate (ATP) | Baseline to 3 months
  A measure of ATP change from baseline to study end
Change in Inorganic Phosphate | Baseline to 3 months
  A measure of inorganic phosphate change from baseline to study end
Change in Phosphodiester | Baseline to 3 months
  A measure of phosphodiester change from baseline to study end
ATPmax production | Baseline to 3 months
  Exercise induced ATPmax production change

SECONDARY OUTCOMES:
Plasma Beta-hydroxybutyrate (β-OH-B) | baseline to 3 months
  Change in β-OH-B with medication
Acetoacetate concentrations | baseline to 3 months
  Change in acetoacetate concentrations
6-min walking test | baseline to 3 months
  Change in the distance that can be covered in a 6 minute walk test
Patient-Reported Outcomes Measure Information System | baseline to 3 months
  By checking KCCQ (Kansas City Cardiomyopathy) scoring: Responses are categorized under 3 sub scales (symptom burden, physical limitation and quality of life) with a range of possible subscale scores from 0 to 100, with 100 representing the least burden of symptoms. The total KCCQ score represents the mean of the three sub scale scores.
plasma ketone concentration on myocardial function | Baseline to 3months + 8 days
  To examine the contribution of the SGLT2i-induced increase in plasma ketone concentration on myocardial function by inhibiting the rise in plasma ketone concentration with acipimox while continuing empagliflozin.
plasma ketone concentration on myocardial blood flow | Baseline to 3months + 8 days
  To examine the contribution of the SGLT2i-induced increase in plasma ketone concentration on myocardial blood flow by inhibiting the rise in plasma ketone concentration with acipimox while continuing empagliflozin.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Texas Diabetes Institute - University Health System, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will actively participate in journal clubs and symposia and present abstracts at national meetings, as well as submit manuscripts to top peer-reviewed journals.
Supporting Information: Study Protocol, SAP